CLINICAL TRIAL: NCT04901286
Title: The Effects of a Single Bout of Moderate Intensity Aerobic Exercise Combined With Different Environments on Executive Function and Processing Speed in Individuals With TBI
Brief Title: The Environment's Impact on Thinking When Added to Leg Cycling in People With TBI: VITAL
Acronym: VITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Carly Wender, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R115220
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Injuries, Traumatic; Aerobic Exercise; Leg Cycling; Virtual Reality
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Exercise

STUDY DESIGN:
Masking Description: The PI will be blinded to the order of conditions for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Seated Rest (No Intervention): Behavioral: Seated Rest In the seated rest control condition, participants will sit on the bike for 30 minutes. Interaction with researchers will be kept at a minimum, similar to that in other sessions. Heart rate will be recorded every two minutes and perceived exertion will be reported every four minutes.
- Exercise Only (Active Comparator): Behavioral: Exercise Only In the exercise-only condition, participants will complete a total of 30-minutes on the stationary bike. This will include a) 5-min warm-up at low resistance, b) 20 minutes of moderate-vigorous intensity cycling, and c) a 5-min cool-down at low resistance. Interaction with researchers will be kept at a minimum, similar to that in other sessions. Heart rate will be recorded every two minutes and perceived exertion will be reported every four minutes.
  Interventions: Behavioral: Exercise Only
- Exercise + Non-Immersive Virtual Reality (Experimental): Behavioral: Exercise + Non-Immersive Virtual Reality In the exercise with non-immersive Virtual Reality condition, participants will complete a total of 30-minutes on the stationary bike while watching a video on an iPad. The cycling session will be identical to that in the Exercise Only condition (5-min warm-up, 20 minutes of moderate-vigorous intensity cycling, and 5-min cool down). During cycling, a YouTube video called "360° VR Cycling Newport Back Bay Sunset [30 MIN - NO MUSIC])" will play on an iPad placed on the front of the bike. Interaction with researchers will be kept at a minimum, similar to that in other sessions. Heart rate will be recorded every two minutes and perceived exertion will be reported every four minutes.
  Interventions: Behavioral: Exercise + Non-Immersive Virtual Reality
- Exercise + Immersive Virtual Reality (Experimental): Behavioral: Exercise + Immersive Virtual Reality In the exercise with immersive virtual reality condition, participants will complete a total of 30-minutes on the stationary bike while wearing Oculus Quest 2 goggles. The bout of cycling will be identical to the prescription given in the exercise only condition (5-min warm-up, 20 minutes of moderate-vigorous intensity cycling, and 5-min cool down). During cycling, the Oculus YouTubeVR app will play a 360° version of the YouTube video called "360° VR Cycling Newport Back Bay Sunset [30 MIN - NO MUSIC])". Interaction with researchers will be kept at a minimum, similar to that in other sessions. Heart Rate will be recorded every two minutes and perceived exertion will be reported every four minutes.
  Interventions: Behavioral: Exercise + Immersive Virtual Reality

INTERVENTIONS:
Behavioral: Exercise Only — Cycling in a lab environment
  Arms: Exercise Only
Behavioral: Exercise + Non-Immersive Virtual Reality — Cycling with an environment simulated by non-immersive virtual reality
  Arms: Exercise + Non-Immersive Virtual Reality
Behavioral: Exercise + Immersive Virtual Reality — Cycling with an environment simulated by immersive virtual reality
  Arms: Exercise + Immersive Virtual Reality

SUMMARY:
Aerobic exercise is a promising treatment modality for cognition in persons with TBI, but effects are consistently small. This study aims to investigate the effect of difference environments during moderate intensity cycling sessions on cognition.

DETAILED DESCRIPTION:
The proposed research study would be the first to investigate the acute effects of aerobic exercise with different environments relative to control and comparison conditions on several domains of cognition in people with TBI. This critical investigation will be a first step toward systematically identifying an optimal exercise training intervention for managing common cognitive consequences of TBI.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age and younger than 59 years of age
* Speak English as their primary language
* Have had a previous TBI at least one year prior\

Exclusion Criteria:

* Have contraindications to moderate or high intensity physical activity, based on the Physical Activity Readiness Questionnaire (PAR-Q)
* Have a history of psychiatric illness (ex: major depression, bipolar disorder, schizophrenia), neurological disorders beyond TBI (ex: stroke, seizure disorder), or substance abuse
* Currently use medications that might impact cognition (ex: steroids, benzodiazepines, neuroleptics)
* Be currently pregnant
* Have visual impairments not otherwise corrected by contact lenses (ex: stereo blindness, colorblindness)
* Have a high likelihood of motion sickness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change on Walking While Talking Test (WWT) | 30 minutes (before and after the acute exercise intervention)
  The WWT measures multitasking by comparing performance on a single motor task to the motor performance during a simultaneous motor + cognitive dual task.
Change on N-Back Test (N-back) | 30 minutes (before and after the acute exercise intervention)
  The N-Back is a measure that requires participants to listen to a sequence of numbers and decide if the current number is the same as the one presented N trials ago.
Change on the Modified Flanker Test (MFT) | 30 minutes (before and after the acute exercise intervention)
  This task requires individuals to correctly respond to a target symbol amid other symbols, ignoring irrelevant information.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No